CLINICAL TRIAL: NCT06224894
Title: The Effect of Music Therapy on Nausea, Vomiting and Anxiety Levels in Children Diagnosed With Oncological Cancer Receiving Cisplatin: Randomized Controlled Study
Brief Title: The Effect of Music Therapy on Nausea, Vomiting and Anxiety Levels in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Principal Investigator, Fulya Kos, lecturer, Bilecik Seyh Edebali Universitesi
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BSEU-HSF
Record Dates: First submitted 2024-01-11; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Music Therapy; Nausea; Anxiety; Cancer; Vomiting; Children, Only
MeSH Terms: conditions — Nausea; Anxiety Disorders; Neoplasms; Vomiting | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music therapy (Experimental): The child in the music therapy group will receive a standard antiemetic treatment procedure 15 minutes before the cisplatin infusion. Music therapy will be applied with the start of cisplatin infusion. The song "The Happiest Child", developed by creating rhythms and developed by Fulya Merve KOS, a researcher with a RhythmotherapistTM certificate issued by the Ministry of National Education, will be used in music therapy. The sound will be adjusted to 45 db. The speaker will be placed at the end of the foot, approximately 30 cm from the child's ear, five minutes before the procedure and will be played to the child during the procedure. After the infusion, music therapy will be terminated and the level of nausea, irritability and anxiety will be evaluated with data collection forms.
  Interventions: Other: Music Therapy; Other: antiemetic treatment
- antiemetic treatment (Experimental): Standard approach; Granisetron IV 40mcg/kg/24, Aprepitant PO 125 mg/24 hour and Dexamethasone 6 mg/m2 IV/PO are administered to children receiving cisplatin treatment.
  Interventions: Other: antiemetic treatment

INTERVENTIONS:
Other: Music Therapy — Music Therapy
  Arms: music therapy
Other: antiemetic treatment — antiemetic treatment

SUMMARY:
This study will be conducted with a randomized controlled study model to examine the effect of music therapy on nausea, vomiting and anxiety levels in children diagnosed with oncological cancer receiving cisplatin.

The research is planned to be carried out at Dokuz Eylül University Nevvar-Salih İşgören Children's Hospital Pediatric Hematology-Oncology Clinic between December 2023 and December 2024. There is no application for music therapy in the operation of this hospital and clinic.

DETAILED DESCRIPTION:
This study was planned to be conducted with children aged 7-18 years old who were hospitalized in the Pediatric Oncology Clinic of Dokuz Eylül University Hospital Nevvar-Salih İşgören Children's Hospital. The sample calculation required for the study was based on a significance level of 0.05, a power of 80% and an effect size of 0.15 (medium effect size) in the GPOWER 3.1 statistical analysis program. It was determined that 33 children should be included in each group for t test analysis in dependent groups. In order to fulfill the parametric test assumptions in the study and considering the 10% loss, it was planned to include 40 children in the experimental group and 40 children in the parent and control group, who voluntarily agreed to participate in the research, for a total of 80 children.

Children with cancer who are between the ages of 7-18, receive cisplatin treatment, are diagnosed with oncological cancer, do not have mental retardation as a clinical diagnosis, receive chemotherapy during their stay in the clinic, have no hearing problems, know how to read and write in Turkish, and volunteer to participate in the study will be included in the study. . Children with cancer who are in the terminal stage and do not want to participate in the study will not be included in the study.

Data Collection Process Children who will receive the intervention and their parents will be informed about the research. Children and their parents will be informed about the music therapy to be applied to their children and their verbal and written consent will be obtained. After consent is obtained, it will be determined which group the child belongs to by randomization method. The standard approach will be applied to all children.

Standard approach; Granisetron IV 40mcg/kg/24, Aprepitant PO 125 mg/24 hour and Dexamethasone 6 mg/m2 IV/PO are administered to children receiving cisplatin treatment.

The child in the control group will not undergo any additional intervention, and the standard antiemetic treatment procedure will be applied 15 minutes before the cisplatin infusion.

The child in the music therapy group will receive a standard antiemetic treatment procedure 15 minutes before the cisplatin infusion. Music therapy will be applied with the start of cisplatin infusion. The song "The Happiest Child", developed by creating rhythms and developed by Fulya Merve KOS, one of the researchers with the RhythmotherapistTM certificate issued by the Ministry of National Education, will be used in music therapy. The sound will be adjusted to 45 db. The speaker will be placed at the end of the foot, approximately 30 cm from the child's ear, five minutes before the procedure and will be played to the child during the procedure. After the infusion, music therapy will be terminated and the level of nausea, irritability and anxiety will be evaluated with data collection forms.

Randomization A total of 80 children who meet the inclusion criteria will be included in the study.

The random selection process of 80 people will be created by the computer randomization program (www.randomizer.org). The Research Randomizer program is a free resource for researchers who need a quick way to generate random numbers or assign participants to experimental conditions. This site may be used for a variety of purposes, including psychology experiments, medical experiments, and survey research.

The program can automatically generate a set of 40 numbers from 1-80 without creating any repetitions. Each child will be randomly assigned a number between 1 and 80. Children given odd numbers will be included in the control group, and children given even numbers will be included in the music therapy group.

ELIGIBILITY:
Example:

Inclusion Criteria:

* Those between the ages of 7-18,
* Receiving Cisplatin Treatment, Diagnosed with Oncological Cancer,
* Without Mental Retardation as a Clinical Diagnosis,
* Those who received chemotherapy during their stay in the clinic,
* No Hearing Problems,
* Able to Read and Write Turkish,
* Children with Cancer who Volunteer to Participate in the Research

Exclusion Criteria:

• Children with cancer who are in the terminal period and do not want to participate in the study will not be included in the study.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
Child and Parent Information Form | one year
  The form, created by the researchers using the literature, consists of 22 questions indicating the child's age, gender, diagnosis, treatment method, medication use other than chemotherapy, medications used, parent's age, parent's education, income and employment status, and characteristics of the child's care and treatment.
Nausea Vomiting Thermometer for Children with Cancer | one year
  It is a visual scale that measures nausea and vomiting developed by Kudubeş and Bektaş in 2022. The scale is thermometer-shaped and has five degrees. It is visualized as a smiling face (1), unresponsive face (2), sad face (3), sad face (4) and crying face (5). Additionally, as the scale score increases, the facial expression on the scale changes. It is scored as never (1), rarely (2), sometimes (3), often (4) and always (5). The lowest score from the scale is 1 and the highest score is 5. An increase in the scale score indicates that the child's degree of nausea and vomiting increases. The intraclass correlation coefficient of the scale is 0.99.
Pediatric Rhodes Nausea and Vomiting Scale Adapted for Children: | one year
  ARINVc was first developed for adult oncology patients by Rhodes and later adapted to children by Lo and Hayman. The validity and reliability study of the scale was conducted by Akçay and his colleagues in the Turkish population in 2018. The scale consists of five statements for each of 6 items measuring the child's frequency, duration and distress of nausea, frequency of vomiting and distress in the last 12 hours and is scored between 0 and 4. ARINVc consists of 6 items. The first three items in the scale question the frequency, amount, and distress caused by vomiting during the last 12 hours, and the remaining three items question the frequency, duration, and distress caused by nausea.
State-Trait Anxiety Scale for Children | one year
  The scale was developed by Spielberger in 1973. Its Turkish validity and reliability was conducted by Özusta in 1995 (Özusta, 1995). In the State Anxiety Scale of ÇDSCI, children are asked to evaluate how they feel 'at that moment' and to mark one of three relevant options. The scale, consisting of 20 items, aims to evaluate emotions related to state anxiety such as tension, irritability, and uneasiness. If the child reports the presence of these feelings as a lot, the highest score is 3, and if the child reports that they do not exist, the lowest score is 1.

IPD SHARING:
Plan to Share IPD: No
no planning